CLINICAL TRIAL: NCT04661748
Title: Continuous Wireless Monitoring of Vital Signs and Automated Alerts of Patient Deterioration vs. Routine Monitoring of High-risk Patients Admitted to Medical Wards
Brief Title: Automated Alerts of Patient Deterioration vs. Routine Monitoring of High-risk Patients Admitted to Medical Wards
Acronym: WARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Katja Kjær Grønbæk, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-20033246
Record Dates: First submitted 2020-12-02; First posted 2020-12-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2023-05

CONDITIONS: Alert Fatigue, Health Personnel; Deterioration, Clinical
MeSH Terms: conditions — Alert Fatigue, Health Personnel; Clinical Deterioration

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): Active alarms
  Interventions: Device: real time alarm of deviating vital signs
- no intervention (No Intervention): No alarms

INTERVENTIONS:
Device: real time alarm of deviating vital signs — Intervention consists of actively alerting staff personnel if physiologic vital signs, deviates from certain thresholds
  Arms: Intervention arm

SUMMARY:
The primary aim of the current study is to assess the effect of continuous wireless vital signs monitoring with generation of real-time alerts compared to blinded monitoring without alerts on the cumulative duration of any severely deviating vital signs in patients admitted to general hospital wards with acute medical conditions. Patients admitted with medical conditions represents a large and heterogenous group occupying a substantial part of the total in-patient capacity in the Danish hospitals today. The hypothesize is that continuous vital signs monitoring, and real-time alerts will reduce the cumulative duration of severely deviating vital signs.

DETAILED DESCRIPTION:
Deterioration of patients on general hospital wards often goes unnoticed for prolonged periods of time. This delay can potentially result in severe adverse outcomes such as cardiopulmonary arrest and need for admission to the intensive care unit (ICU). These complications occur despite the fact that, in most cases, measurable changes in physiological vital signs, could identify patients at risk. Moreover, occurrence of complications increase treatment costs considerably underpinning the rationale of early detection of patient deterioration in both human and economic terms.

Monitoring of vital signs outside of ICU or telemetry units usually relies on intermittent manual assessments performed by clinical staff at intervals of up to 12 hours with the "Early Warning Score (EWS)", "Tidlig Opsporing af Kritisk Sygdom (TOKS)" or similar systems. However, significant deterioration may occur in-between these intervals, which may explain the EWS/TOKS score's proven lack of impact on morbidity and mortality in Danish hospitals.

Recent medico-technical advances have allowed for clinical use of small wireless wear-and-forget devices that continuously monitor various indices of cardiopulmonary status, ambulatory activity, temperature etc. Studies suggest that integration of continuous monitoring into automated patient surveillance systems more often detects cardiorespiratory instability and may decrease number of Emergency Response Team activations, ICU transfers, length of hospital stay, morbidity and mortality but further randomized controlled trials (RCTs) are needed to confirm this. Other advantages may be a decrease in the time required for vital signs measurement and recording compared to routine monitoring and overall health care cost savings with return-on-investment estimates ranging from 127%-1739%.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion and randomization possible within 12 hours of fulfilling all other inclusion criteria below.
* Adult patients (≥18 years).
* At least one (additional) expected overnight stay.
* High-risk medical admission, defines as EITHER:

  * one or more of the following symptoms or tentative diagnoses: Pneumonia, dyspnea, acute coronary syndrome, new onset heart failure or sepsis WITH two or more of the following deviations in vital signs recorded at one time point within 48 hours of admission:

    * Respiratory rate ≥ 21 min-1 or ≤ 7 min-1
    * Oxygen saturation of arterial hemoglobin ≤ 93 %
    * Pulse rate ≥ 111 min-1 or ≤ 40 min-1
    * Systolic blood pressure ≤ 100 mmHg or > 200 mmHg
    * Temperature > 39 °C or ≤ 35,9 °C
    * Any alteration in mental status
    * Any oxygen supplementation

OR

○ Discharged from ICU-stay lasting ≥ 24 hours regardless of cause of ICU-admission.

Exclusion Criteria:

* Patient expected not to cooperate with study procedures.
* Allergy to plaster or silicone.
* Patients admitted for palliative care only (i.e. no active treatment).
* Planned admission to unit using continuous vital sign monitoring (i.e. an intermediary care/telemetry unit).
* Patients previously enrolled in the studies WARD-COPD (H-18026653) or WARD-Surgery (H-17033535).
* Patients previously enrolled in the surgical ward RCT
* A pacemaker or Implantable Cardioverter Defibrillator (ICD) device.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative duration of one or more of the following deviations in vital signs during the first five days of admission or until discharge: | 5 days after inclusion or until discharge
  ● SpO2 < 85%
Cumulative duration of one or more of the following deviations in vital signs during the first five days of admission or until discharge: | 5 days after inclusion or until discharge
  * Respiratory rate ≤ 5 min-1
  * Respiratory rate > 24 min-1
Cumulative duration of one or more of the following deviations in vital signs during the first five days of admission or until discharge: | 5 days after inclusion or until discharge
  * Heart rate > 130 min-1
  * Heart rate ≤ 30 min-1
Cumulative duration of one or more of the following deviations in vital signs during the first five days of admission or until discharge: | 5 days after inclusion or until discharge
  * Systolic blood pressure ≤ 90 mmHg
  * Systolic blood pressure > 220 mmHg
Cumulative duration of one or more of the following deviations in vital signs during the first five days of admission or until discharge: | 5 days after inclusion or until discharge
  ● Atrial fibrillation
Cumulative duration of one or more of the following deviations in vital signs during the first five days of admission or until discharge: | 5 days after inclusion or until discharge
  ● Circulatory failure
  * Systolic blood pressure < 100 mmHg AND
  * Heart rate >110 min-1 (for more than 30 minutes) OR heart rate >130 min-1 (for more than 5 minutes) OR heart rate < 50 (for more than 30 minutes) AND/

SECONDARY OUTCOMES:
Frequency and duration of deviations in vital signs | 5 days after inclusion or until discharge
  Frequency of each of the deviations in vital signs. List of vital signs, and normal limits detailed in protocol

OTHER OUTCOMES:
Number of patients with any adverse clinical outcomes | 30 days after inclusion
  Any adverse events. Criteria for each defined in protocol. Adverse events will be manually categorised as a 'Severe adverse event' (SAE), or simple 'adverse event' (AE).
Length of hospital stay (LOS) | 6 months after inclusion
  Lenght of hospital stay
Total patient-related healthcare expenses in patients experiencing adverse clinical outcomes compared to patients without such outcomes and the effect of the study intervention on expenses | 2 years
  Total patient-related healthcare expenses in patients experiencing adverse clinical outcomes compared to patients without such outcomes and the effect of the study intervention on expenses
Staff response time (interventions group only) | 5 days after inclusion
  Time from the staff is notified by app, until they respond by selecting 'check on patient' in app Stratified according to time of day

CONTACTS AND LOCATIONS:
Overall Officials: Katja K Grønbæk, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg and Frederiksberg Hospital, København NV, Region H, Denmark

IPD SHARING:
Plan to Share IPD: Undecided